CLINICAL TRIAL: NCT05411796
Title: In-Use Randomized, Cross-over, Double-blind Study of Two Different Menstrual Cups
Brief Title: In-use Cross-over Study of Two Different Menstrual Cups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CSD 2018094
Record Dates: First submitted 2022-05-20; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Menstruation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: menstrual cups distributed in unmarked packaging; participants and investigator blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tampax menstrual cup (regular flow), then Other menstrual cup (size 1) (Experimental)
  Interventions: Device: Tampax menstrual cup; Device: Other menstrual cup
- Other menstrual cup (size 1), then Tampax menstrual cup (regular flow) (Experimental)
  Interventions: Device: Tampax menstrual cup; Device: Other menstrual cup

INTERVENTIONS:
Device: Tampax menstrual cup — regular flow size
Device: Other menstrual cup — size 1

SUMMARY:
This study evaluated the safety and tolerability of two different menstrual cups on vaginal health

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrollment into this study subjects must meet the following criteria (i.e., responses = "Yes"):

1. Have you read, understood, and signed the Informed Consent?
2. Have you read, understood and signed the Confidentiality Agreement?
3. Are you female, between 18 and 55 years of age (inclusive)?
4. For at least the last 4 months, have you had a consistent monthly menstrual cycle lasting 21-35 days with menstrual bleeding lasting at least 3 days' duration?
5. Are you willing to wear the cup at least 12 hours (may remove to empty) a day and a minimum of 3 days during your menstrual cycle?
6. Do you agree to use at least one form of birth control (i.e., intrauterine device, oral contraceptives, contractive implants or injections, diaphragm with spermicide, cervical cap, tubal ligation, partner had vasectomy or use of condom) if you are of child-bearing potential for the duration of the study? Note: Abstinence will be considered birth control in women not sexually active
7. Do you primarily use tampons (no slim/ultra slim) or menstrual cup for your feminine protection needs during your periods (may use pads and/or pantiliners as back-up/overnight use)?
8. Is your typical menstrual flow moderate/medium, heavy or extra heavy?
9. Do you wear tampons or menstrual cups during menstruation with no abnormal discomfort?
10. Was your last Papanicolaou (PAP) smear normal in the past 3 years (or have a normal PAP with a negative Human Papilloma Virus (HPV) in the past 5 years)? NOTE: Women age 18-20 do NOT need a PAP regardless of sexual activity or not (per ACOG guidelines), (self-reported)
11. In the past 48 hours, have you refrained from - and do you agree to continue to refrain from - vaginal intercourse within the 48 hours before each visit?
12. Have you refrained from showering within 12 hours and/or bathing within 24 hours of this visit - and do you agree to continue to refrain from - showering within 12 hours and/or bathing within 24 hours before each visit?
13. In the past 48 hours, have you refrained from - and do you agree to continue to refrain from - using douching substances, feminine hygiene products, powders, perfumes, wipes, lotions, creams, or emollients to your genital area for the duration of the study?
14. Do you agree to refrain from genital hair removal (e.g. waxing, shaving, etc.) while on the study?
15. Do you agree to refrain from using antibacterial body soap while on the study? NOTE: Hand washing is ok (e.g., Safeguard®, Dial®)
16. Have you refrained from - and do you agree to continue to refrain from - using antihistamines (e.g., Benadryl®) or non-steroidal anti-inflammatory medication (e.g. Advil®, Aspirin) for at least 3 days prior to each visit?
17. Do you agree to refrain from participation in other concurrent clinical research studies?
18. Do you agree to only use the menstrual cups, pads and pantiliners supplied at each study visit for menstrual protection while participating in this study?
19. Do you agree to refrain from using tampons during this study?
20. Do you agree to complete all study questionnaires and diaries?
21. Are you willing to keep fingernails at a suitable length and condition to help prevent injury during product insertion and removal?
22. Are you willing and able to comply with the study requirements?
23. SITE: Is the subject in generally good health? (without clinically significant disease as determined by Investigator/Designee based on medical history and vaginal exam)

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following (i.e., responses = "Yes"):

1. Have you had a menstrual abnormality with any of your last menstrual cycles in the last 4 months (such as oligomenorrhea or amenorrhea, or bleed more than 7 days a month)?
2. Have you had a vaginal delivery in the last 6 months?
3. Are you pregnant (SITE: per urine pregnancy test at screening), lactating or planning to become pregnant during the duration of the study?
4. Have you had vaginal surgery, perineal surgery, uterine surgery, miscarriage or abortion (spontaneous or induced) in the last 6 months?
5. Do you have difficulty emptying your bladder?
6. Do you have a history of Toxic Shock Syndrome (TSS)?
7. Have you taken steroids within the past seven days? Exception: Topical steroids outside the perineal/vaginal area are okay, at the discretion of the Investigator.
8. Do you currently or have you taken anticoagulants within the last 30 days (e.g., Coumadin® [warfarin], Eliquis® and/or Xarelto®) or have a bleeding disorder? (self-reported)?
9. Do you have a vulvar piercing?
10. Do you have a history of genital herpes?
11. Within the last 6 months have you had endometrial disease/uterine fibroids with heavy menstrual flow?
12. Have you been diagnosed or had a chemical dependence within the last 2 years (e.g., opiates, marijuana, etc.)? (self-reported).
13. Do you currently have a urinary tract infection (UTI) or a history of frequent UTIs (> 2 times within previous 12 months)? (self-reported).
14. Do you have urinary incontinence which causes you to regularly use and saturate diapers or absorbent panties or pads (more than 3 times a week over the last 4 months), or have you been treated for a pelvic floor disorder (e.g., perineal floor re-education with vaginal probe) within last 6 months?
15. Are you currently using a vaginal probiotic therapy? (self-reported).
16. Have you participated in a clinical study with exposure to any investigational product within the last 30 days?
17. Have you taken any antibiotics or antifungals within last 4 weeks? Note: Topical use of antibiotics or antifungals outside the perineal/genitourinary area is allowed at the discretion of the Investigator.
18. Have you started a new hormonal birth control in the last 4 months, or plan changing hormonal birth control during the study period?
19. Do you have a history of Light Emitting Diode(LED) or laser vaginal therapy within the last 6 months? (self-reported).
20. Are you or a household member employed by any subsidiaries in the feminine care or incontinence business, including Procter & Gamble, Johnson & Johnson, Kimberly Clark, Energizer Holdings, SCA, Unicharm, Diva Cup International and First Quality?
21. SITE: Has the subject been diagnosed with a medical condition which might compromise the immune system including cancer, anemia, blood disorders, or malnutrition within the last 2 years? Exception - Successfully removed non-melanoma skin cancers outside the test area are okay at the discretion of the Investigator (self-reported).
22. SITE: Does the subject have uncontrolled and/or unstable diabetes in the opinion of the Investigator? Note: Must be on stable dose of medication for at least 6 months.
23. SITE: Does the subject have a history of immunosuppressive drug therapy, chemotherapy, or radiation therapy?
24. SITE: Does the subject have history of or current diagnosis of AIDS/HIV, organ transplant, liver disease, renal disease, deep vein thrombosis, pulmonary embolism, haemophilia, autoimmune disease, thyroid disorder, major depression, Crohn's disease, Irritable Bowel Disease or any other medical condition, which in the opinion of the Investigator would preclude study participation? Note: For thyroid: acceptable if on a stable dose of medication for at least 6 months.
25. SITE: Does the subject have a vaginal erythema grade of > 2 or a score of > 1.0 for abrasions, ulcerations and/or lacerations as determined by the Investigator at the screening visit?
26. SITE: Has the subject been diagnosed with an atrophic vagina defined as thin, friable vaginal epithelium that bleeds on speculum examination (i.e. undiagnosed atrophy; subject may report experiencing pain on intercourse) (self-reported)?
27. SITE: Has the subject been diagnosed with pelvic organ prolapse in any compartment (anterior, apical or posterior)?
28. SITE: Does the subject have active vaginal infections (Chlamydia trachomatis and/or Neisseria gonorrhoeae) identified through lab results from the microbiological sample obtained at the screening visit?
29. SITE: Does the subject have active genital warts, lesions, and/or vaginal infections (such as bacterial vaginosis (BV), Candida spp., Trichomonas vaginalis) at the screening visit?

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females with regular menstrual cycles
Enrollment: 65 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Vaginal erythema | within 72 hours of last menstrual cup use
  visually graded on a scale of 0 (no apparent erythema) to 4 (severe erythema)

SECONDARY OUTCOMES:
Vaginal abrasion | within 72 hours of last menstrual cup use
  visually graded on a scale of 0 (intact) to 2 (deep disruption)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Noss, M.D., Principal Investigator — Synexus, Inc
Locations (1):
- Synexus-US, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No